CLINICAL TRIAL: NCT03597386
Title: ConfirmMDx Assay is Multiparametric MRI (mpMRI) PIRADS Scored Lesions After a Negative MR/US Fusion Biopsy
Brief Title: ConfirmMDx Assay in Multiparametric MRI (mpMRI) PIRADS Scored Lesions After a Negative MR/US Fusion Biopsy
Status: Withdrawn | Type: Observational
Why Stopped: The study will not be conducted
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Hani Rashid, Professor, Urology, University of Rochester
Other Study IDs: 71689
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Prostate Disease
MeSH Terms: conditions — Prostatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — MR/US prostate fusion biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants

SUMMARY:
The purpose of this study is to see if the ConfirmMDx assay is useful in finding prostate cancer in patients who are at increased risk for prostate cancer based on elevated PSA and prostate lesion identified on mpMRI.

ELIGIBILITY:
Inclusion Criteria:

* Prior documented elevated PSA (> 4.0 ng/ml)
* MRI lesion based on PIRADS scoring within the past 3 years
* Completed MR/US fusion prostate biopsy with concurrent systematic biopsy for PIRADS score 2-5 with negative pathological findings completed subsequent ConfirmMDx assay (regardless of result). The most recent biopsy can be within 4 years if ConfirmMDx already completed.
* May have had prior negative biopsy sessions prior to the most recent MR/US fusion biopsy
* Must be able to stop anticoagulation/antiplatelet therapy 5-7 days prior to obtaining biopsy
* Ability to give informed consent

Exclusion Criteria:

* Any metastatic cancer
* Any prostate cancer
* Active infection: urinary tract infection or prostate infection precluding prostate biopsy
* Anal stenosis or severe anal disease preventing prostate biopsy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men are eligible for this prostate study
Study Population: Subjects were selected due to increased risk of prostate cancer with prior elevated prostate specific antigen (PSA), mpMRI, prostatic lesions and negative MRI-ultrasound guided fusion biopsy due to the potential for prostate cancer that was not detected prior.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Detection of prostate cancer based on rebiopsy of lesions on multiparametric MRI (mpMRI) following a negative MR/US fusion biopsy with concurrent systematic biopsy with correlation of ConfirmMDx assay testing performed on negative MR/US fusion biopsy | baseline

SECONDARY OUTCOMES:
Correlation of PIRADS scores with ConfirmMDx testing outcomes | baseline
Correlation of prostate cancer detection on re-biopsy with ConfirmMDx testing outcomes | baseline
Compare prostate cancer detection rates for repeat MR/US fusion biopsy after prior negative biopsy | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No